CLINICAL TRIAL: NCT05455359
Title: The Impact of Upper Gastrointestinal Dysmotility on Aspiration-associated Symptoms
Brief Title: Gastrointestinal Dysmotility on Aspiration Risk
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Rachel Rosen, Associate Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-P00038381
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Motility Disorders; Gastric Motor Dysfunction; Aspiration Pneumonia; Gastro Esophageal Reflux
MeSH Terms: conditions — Esophageal Motility Disorders; Pneumonia, Aspiration; Gastroesophageal Reflux | interventions — prucalopride; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Patients will be undergo 1 week observation period followed by 4 weeks of prucalopride followed by 1 weeks of a wash out followed by 4 weeks of famotidine
  Interventions: Drug: Prucalopride; Drug: Famotidine
- Arm 2 (Experimental): Patients will be undergo 1 week observation period followed by 4 weeks of famotidine followed by 1 weeks of a wash out followed by 4 weeks of prucalopride
  Interventions: Drug: Prucalopride; Drug: Famotidine

INTERVENTIONS:
Drug: Prucalopride — Prucalopride 0.04 mg/kg/day
Drug: Famotidine — Famotidine 0.4 mg/kg/day

SUMMARY:
The hypothesis of this study is that esophageal and gastric dysmotility increase the risk of developing aspiration-associated symptoms in children with neurologic impairment. The investigators are conducting a ten week cross over study comparing prucalopride to famotidine for the treatment of aspiration-associated symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. are 5-21 years of age;
2. receive >90% of their calories by enteral tube (i.e., patients take no food or drink by mouth);
3. are determined to be at high risk for aspiration pneumonia based on evidence of impaired airway protective mechanisms, documented by aspiration on video fluoroscopic swallow study;
4. have static neurologic impairment, defined as functional and/or intellectual impairment that results from a chronic neurologic or related diagnosis (e.g., cerebral palsy) with no prospect of progression for at least one year;
5. have chronic respiratory symptoms, defined as coughing, choking, or need for oral suctioning a minimum of three times per week during the prior four weeks.

   -

Exclusion Criteria:

1. have progressive neurologic impairment;
2. have a history of prior intact Nissen fundoplication;
3. are currently taking oral or inhaled antibiotics, including prophylactic antibiotics;
4. are currently taking or have taken in the last four weeks acid suppression (H2 antagonist or PPI); or
5. are fed by gastrojejunostomy rather than by gastrostomy. -

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Pediatric Cough Quality of Life Questionnaire | 4 weeks
  Comparison of the mean difference in the Pediatric Cough Quality of Life Questionnaire (range: 7 to 189, lower scores=more symptom impairment) between baseline and 4 week scores between Arm 1 and Arm 2

SECONDARY OUTCOMES:
Gastric emptying outcomes | 4 weeks
  Comparison of within-patient differences in gastric residuals by nuclear scintigraphy
Total Peds-GI QL score | 8 weeks
  Comparison of the mean difference in total Peds-GI QL scores (range: 0-100, lower=worse symptoms) between famotidine and prucalopride periods
Aspiration symptoms | 4 weeks
  Comparison of the mean difference in the number of coughing or choking episodes per week during the fourth week of treatment
Microbiome | 8 weeks
  Comparison of within-patient differences in microbiome diversity and abundance between baseline and after each medication period
Pneumonias | 10 weeks
  Comparisons in the number of aspiration pneumonias between each treatment period
Esophageal reflux events | 4 weeks
  Comparison of within-patient differences in post-prandial reflux events by nuclear scintigraphy

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No